CLINICAL TRIAL: NCT06492525
Title: A Phase 1, Open-label, 2-period, Fixed Sequence, Cross-over Study To Investigate The Effect Of Multiple Doses Of Rifampicin Or Itraconazole On The Pharmacokinetics Of Single Dose Ensartinib In Healthy Volunteers.
Brief Title: A Study To Evaluate The Effect Of Rifampicin Or Ltraconazole On Pharmacokinetics Of Ensartinib In Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BTP-42319
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — ensartinib; Rifampin; Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): All subjects in this cohort will receive the same dose of Ensartinib in both periods. Subjects will receive Ensartinib Alone in Period 1 followed by Ensartinib with Rifampicin in Period 2.
  Interventions: Drug: Ensartinib; Drug: Rifampicin
- Cohort 2 (Experimental): All subjects in this cohort will receive the same dose of Ensartinib in both periods. Subjects will receive Ensartinib Alone in Period 1 followed by Ensartinib with Itraconazole in Period 2.
  Interventions: Drug: Itraconazole; Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — 225 mg oral dose on day 1 in period 1 and on day 18 in period 2
  Arms: Cohort 1
Drug: Rifampicin — 600 mg QD from day 9 to day 22 in period 2
  Arms: Cohort 1
Drug: Itraconazole — 200 mg QD from day 9 to day 19 in period 2
  Arms: Cohort 2
Drug: Ensartinib — 100 mg oral dose on day 1 in period 1 and on day 12 in period 2
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to estimate the effect of rifampicin or itraconazole on the single dose PK of ensartinib.

ELIGIBILITY:
Inclusion Criteria:

* Male body weight ≥ 50kg, female body weight ≥ 45kg, body mass index (BMI) within the range of 19 ~ 26kg /m2;
* Clinical laboratory evaluations within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator;
* The subjects should took effective contraceptive measures voluntarily from informed consent until 3 months after Study Completion；
* Able to comprehend and willing to sign an informed consent form.

Exclusion Criteria:

* Those with a history of chronic systemic or serious diseases such as cardiovascular, liver, kidney, lung, gastrointestinal, nervous, musculoskeletal, hematopoietic or metabolic diseases, especially surgical conditions or conditions that may affect drug absorption, distribution, metabolism and excretion；
* Family history or presence of long QTc syndrome; History or presence of an abnormal ECG；
* Hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), treponema pallidum antibody or human immunodeficiency virus antigen/antibody (HIV-Ag/Ab) is positive；
* Use of any medications (prescription drugs, over-the-counter drugs, Chinese herbal medicines, health products, moderate or strong CYP3A inhibitors or inducers, etc) within 14 days prior to the first administration；
* Those who have special dietary requirements (habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeinated beverages) and are unable to withdraw during the trial；
* Drug abusers, smokers or alcoholics；
* Those with a history of fear of needles and hemophobia, difficulty in blood collection or inability to tolerate venipuncture blood collection;
* Donation of blood ≥ 400 mL or receipt of blood products within 3 months before enrollment;
* Receive any vaccine within 1 months before enrollment；
* Participation in any other investigational drug study within 3 months before enrollment；
* History of significant hypersensitivity to any drug compound or food；
* Other conditions that, in the opinion of the investigator, are not suitable for the subject to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Plasma AUC0-t for Ensartinib Given Alone and With Rifampicin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose on Day 1 after Ensartinib 225 mg administration in Period 1, and at the same time points on Day 18 after Ensartinib 225 mg with rifampin administration in Period 2.
  AUC0-t is the plasma area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (Clast).
Plasma AUC0-t for Ensartinib Given Alone and With Itraconazole | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post-dose on Day 1 after Ensartinib 100 mg administration in Period 1, and at the same time points on Day 12 after Ensartinib 100 mg with Itraconazole administration in Period 2.
  AUC0-t is the plasma area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (Clast).
Plasma AUC0-∞ for Ensartinib Given Alone and With Rifampicin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose on Day 1 after Ensartinib 225 mg administration in Period 1, and at the same time points on Day 18 after Ensartinib 225 mg with rifampin administration in Period 2.
  AUC0-∞ is the plasma area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Plasma AUC0-∞ for Ensartinib Given Alone and With Itraconazole | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post-dose on Day 1 after Ensartinib 100 mg administration in Period 1, and at the same time points on Day 12 after Ensartinib 100 mg with Itraconazole administration in Period 2.
  AUC0-∞ is the plasma area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Plasma Cmax for Ensartinib Given Alone and With Rifampicin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose on Day 1 after Ensartinib 225 mg administration in Period 1, and at the same time points on Day 18 after Ensartinib 225 mg with rifampin administration in Period 2.
  Maximum plasma concentration
Plasma Cmax for Ensartinib Given Alone and With Itraconazole | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post-dose on Day 1 after Ensartinib 100 mg administration in Period 1, and at the same time points on Day 12 after Ensartinib 100 mg with Itraconazole administration in Period 2.
  Maximum plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No